CLINICAL TRIAL: NCT00005436
Title: Lupus Cohort--Thrombotic Events and Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4364; R29HL047080 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Thrombosis; Heart Diseases; Lupus Erythematosus, Systemic
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Thrombosis; Heart Diseases; Lupus Erythematosus, Systemic

SUMMARY:
To study longitudinally the incidence, pathogenesis, and risk factors for thrombotic events and coronary artery disease in a cohort of patients with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
BACKGROUND:

The Johns Hopkins Lupus Cohort, begun by Dr. Petri in 1987, was a longitudinal study of the incidence and pathogenesis of thrombotic events and coronary artery disease in SLE. The usual natural history of thrombotic events and coronary artery disease is telescoped in SLE, so that patients present with these outcomes in their third and fourth decades.

DESIGN NARRATIVE:

Risk factors addressed in the study included: 1) the hypercoagulable state secondary to antiphospholipid antibodies (the lupus anticoagulant and anticardiolipin antibody); 2) premature atherosclerosis, accelerated by prednisone and hypertension; 3) underlying vascular damage from lupus vasculopathy and vasculitis; 4) co-morbid factors, including obesity, smoking, hyperlipidemia, hypertension, sedentary life style, and family history of coronary artery disease, and 5) other factors, including sex, age, race, immunogenetics, compliance with medication, and socioeconomic status. The Hopkins Cohort Study was uniquely able to focus on these issues, both because of its population, which reflected a broad racial, educational, and socioeconomic background, and because the four years of data accumulated showed promising preliminary results.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-09; Study Completion 1996-08 (Actual)

REFERENCES:
- [Background] Petri M. Antiphospholipid antibody syndrome: an acquired cause of venous and arterial hypercoagulability. Mt Sinai J Med. 1997 Nov;64(6):376-82. PMID 9364831
- [Background] Bluemke DA, Petri M, Zerhouni EA. Femoral head perfusion and composition: MR imaging and spectroscopic evaluation of patients with systemic lupus erythematosus and at risk for avascular necrosis. Radiology. 1995 Nov;197(2):433-8. doi: 10.1148/radiology.197.2.7480688.
- [Background] Petri M, Robinson C. Oral contraceptives and systemic lupus erythematosus. Arthritis Rheum. 1997 May;40(5):797-803. doi: 10.1002/art.1780400504. PMID 9153538
- [Background] Dunn JP, Noorily SW, Petri M, Finkelstein D, Rosenbaum JT, Jabs DA. Antiphospholipid antibodies and retinal vascular disease. Lupus. 1996 Aug;5(4):313-22. doi: 10.1177/096120339600500413. PMID 8869905
- [Background] Petri M. Hopkins Lupus Pregnancy Center: 1987 to 1996. Rheum Dis Clin North Am. 1997 Feb;23(1):1-13. doi: 10.1016/s0889-857x(05)70311-2. PMID 9031371
- [Background] Sullivan KE, Wisnieski JJ, Winkelstein JA, Louie J, Sachs E, Choi R, Veksler E, Goldman D, Petri M. Serum complement determinations in patients with quiescent systemic lupus erythematosus. J Rheumatol. 1996 Dec;23(12):2063-7. PMID 8970042
- [Background] Petri M. Pathogenesis and treatment of the antiphospholipid antibody syndrome. Med Clin North Am. 1997 Jan;81(1):151-77. doi: 10.1016/s0025-7125(05)70509-5. PMID 9012759
- [Background] Sullivan KE, Wooten C, Goldman D, Petri M. Mannose-binding protein genetic polymorphisms in black patients with systemic lupus erythematosus. Arthritis Rheum. 1996 Dec;39(12):2046-51. doi: 10.1002/art.1780391214. PMID 8961910
- [Background] Petri M, Roubenoff R, Dallal GE, Nadeau MR, Selhub J, Rosenberg IH. Plasma homocysteine as a risk factor for atherothrombotic events in systemic lupus erythematosus. Lancet. 1996 Oct 26;348(9035):1120-4. doi: 10.1016/S0140-6736(96)03032-2. PMID 8888164
- [Background] Petri M. Hydroxychloroquine use in the Baltimore Lupus Cohort: effects on lipids, glucose and thrombosis. Lupus. 1996 Jun;5 Suppl 1:S16-22. PMID 8803905
- [Background] Petri M, Ho AC, Patel J, Demers D, Joseph JM, Goldman D. Elevation of maternal alpha-fetoprotein in systemic lupus erythematosus: a controlled study. J Rheumatol. 1995 Jul;22(7):1365-8. PMID 7562773
- [Background] Mont MA, Glueck CJ, Pacheco IH, Wang P, Hungerford DS, Petri M. Risk factors for osteonecrosis in systemic lupus erythematosus. J Rheumatol. 1997 Apr;24(4):654-62. PMID 9101497
- [Background] Casciola-Rosen L, Rosen A, Petri M, Schlissel M. Surface blebs on apoptotic cells are sites of enhanced procoagulant activity: implications for coagulation events and antigenic spread in systemic lupus erythematosus. Proc Natl Acad Sci U S A. 1996 Feb 20;93(4):1624-9. doi: 10.1073/pnas.93.4.1624. PMID 8643681
- [Background] Petri M. Musculoskeletal complications of systemic lupus erythematosus in the Hopkins Lupus Cohort: an update. Arthritis Care Res. 1995 Sep;8(3):137-45. doi: 10.1002/art.1790080305. PMID 7654797
- [Background] Johnson MJ, Petri M, Witter FR, Repke JT. Evaluation of preterm delivery in a systemic lupus erythematosus pregnancy clinic. Obstet Gynecol. 1995 Sep;86(3):396-9. doi: 10.1016/0029-7844(95)00186-U. PMID 7651650
- [Background] Bermas BL, Petri M, Goldman D, Mittleman B, Miller MW, Stocks NI, Via CS, Shearer GM. T helper cell dysfunction in systemic lupus erythematosus (SLE): relation to disease activity. J Clin Immunol. 1994 May;14(3):169-77. doi: 10.1007/BF01533366. PMID 7929693
- [Background] Bermas BL, Petri M, Berzofsky JA, Waisman A, Shearer GM, Mozes E. Binding of glycoprotein 120 and peptides from the HIV-1 envelope by autoantibodies in mice with experimentally induced systemic lupus erythematosus and in patients with the disease. AIDS Res Hum Retroviruses. 1994 Sep;10(9):1071-7. doi: 10.1089/aid.1994.10.1071. PMID 7826694
- [Background] Petri M, Lakatta C, Magder L, Goldman D. Effect of prednisone and hydroxychloroquine on coronary artery disease risk factors in systemic lupus erythematosus: a longitudinal data analysis. Am J Med. 1994 Mar;96(3):254-9. doi: 10.1016/0002-9343(94)90151-1. PMID 8154514
- [Background] Utset TO, Golden M, Siberry G, Kiri N, Crum RM, Petri M. Depressive symptoms in patients with systemic lupus erythematosus: association with central nervous system lupus and Sjogren's syndrome. J Rheumatol. 1994 Nov;21(11):2039-45. PMID 7869307
- [Background] Watson RM, Scheel JN, Petri M, Kan JS, Provost TT, Ratrie H 3rd, Callan NA. Neonatal lupus erythematosus. Report of serological and immunogenetic studies in twins discordant for congenital heart block. Br J Dermatol. 1994 Mar;130(3):342-8. doi: 10.1111/j.1365-2133.1994.tb02931.x. PMID 8148276
- [Background] Petri M, Watson R, Winkelstein JA, McLean RH. Clinical expression of systemic lupus erythematosus in patients with C4A deficiency. Medicine (Baltimore). 1993 Jul;72(4):236-44. doi: 10.1097/00005792-199307000-00003. PMID 8341140
- [Background] Petri M, Allbritton J. Fetal outcome of lupus pregnancy: a retrospective case-control study of the Hopkins Lupus Cohort. J Rheumatol. 1993 Apr;20(4):650-6. PMID 8496859
- [Background] Petri M. Systemic lupus erythematosus and pregnancy. Rheum Dis Clin North Am. 1994 Feb;20(1):87-118. PMID 8153405